CLINICAL TRIAL: NCT03246802
Title: High Dose Rate Partial Prostate Brachytherapy as Salvage Treatment for Local Failures After Previous External Beam Radiotherapy
Brief Title: Partial Prostate Salvage High Dose Rate Brachytherapy
Acronym: SalvageHDR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Juanita Crook, Professor of Radiation Oncology, British Columbia Cancer Agency
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H17-01641
Record Dates: First submitted 2017-08-03; First posted 2017-08-11 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Prostate Cancer
Keywords: recurrent prostate cancer; mpMRI; salvage HDR brachytherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: High Dose Rate brachytherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HDR partial prostate brachytherapy (Experimental): 2 fractions of high dose rate prostate brachytherapy will be delivered to the site of recurrent disease as determined by mp-MRI
  Interventions: Radiation: HDR partial prostate brachytherapy

INTERVENTIONS:
Radiation: HDR partial prostate brachytherapy — temporary radioactive implant

SUMMARY:
A dose-response relationship for radiation in the management of prostate cancer is well established. Local recurrence of prostate cancer after external beam radiotherapy occurs in at least 40% of patients treated because of inability to deliver sufficient dose through external beam techniques. These patients respond well to re-irradiation using brachytherapy with about 50% of selected patients remaining free of recurrence 5 years after salvage. Advanced imaging using multiparametric Magnetic Resonance Imaging (mpMRI) allows identification of the site of recurrence, permitting partial prostate salvage brachytherapy. There is extensive literature on Low Dose Rate salvage brachytherapy but less on High Dose Rate.

DETAILED DESCRIPTION:
Appropriately selected patients with histologically documented recurrence 3 years or more after initial external beam radiotherapy will undergo mpMRI for identification of the site of recurrence. A planning transrectal ultrasound (TRUS) will be obtained for fusion with the mpMRI and transposition of the target volume (GTV=gross tumor volume). A margin of 4.5 cm will be added to the GTV to create a focal planning target volume (PTV). The margin may be cropped at the interface with critical organs. Two fractions of HDR brachytherapy will be delivered, each from a single implant, 2 weeks apart. Following treatment patients will be monitored for toxicity and quality of life using the Expanded Prostate cancer Index (EPIC) questionnaire as well as the International Prostate Symptom score. Efficacy will be evaluated by monitoring the Prostate Specific Antigen (PSA) and repeat mpMRI at 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >45 and Life expectancy >10 years
* Previous External Beam Radiotherapy (EBRT) dose up to 78Gray/39 fractions, 81 Gray/45 fractions or 70 Gray/28 fractions or LDR brachytherapy with site of recurrence in an under-dosed or untreated site
* > 3 year interval since EBRT or LDR Brachytherapy
* No late toxicity from prior EBRT ≥ grade 2
* Rising PSA post EBRT > nadir + 2 ng/ml but < 10 ng/ml
* PSA Doubling time > 6 months
* Negative staging with CT scan of the abdomen/pelvis and bone scan (PSMA PET scan can replace CT and bone scan)
* Able to undergo multiparametric MRI with endorectal coil
* Radiographic evidence of dominant intraprostatic lesion (DIL) as only area of recurrence (i.e unifocal recurrence) and corresponding to site of original disease
* Biopsy confirmation of DIL with pathology review by British Columbia Cancer Agency GenitoUrinary pathologist (TB)
* Willing to provide informed consent
* History and physical examination within 90 days of registration
* ECOG performance status 0-1 prior to registration
* IPSS < 16, or adequate voiding study (post void residual < 100cc and peak flow rate > 10 cc/second).
* No prior trans urethral prostatic resection
* Recurrence suitable for implant with HDR brachytherapy as assessed on ultrasound simulation (maximum PTV ideally < 65% of prostate volume)
* No history of inflammatory bowel disease or previous rectal surgery
* Suitable for procedure under anesthesia, spinal or general
* INR <2.5 and platelet count >75 x 109/L
* Androgen Deprivation Therapy may be initiated at the discretion of the treating oncologist

Exclusion Criteria:

* Not compliant with criteria above
* Unable to give informed consent

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2032-01-01 (Estimated); Study Completion 2037-01-01 (Estimated)

PRIMARY OUTCOMES:
Late adverse gastrointestinal or genitourinary events grade 3 or higher | 3-60 months
  Common Terminology Criteria for Adverse Events (CTCAE V4.0)

SECONDARY OUTCOMES:
Late Quality of Life | 3-60 months
  Expanded Prostate Cancer Index (EPIC)
Late lower urinary tract symptoms | 3-60 months
  International Prostate Symptom Score
Acute grade 3 or higher gastrointestinal or genitourinary adverse events | 0-3 months
  Common Terminology Criteria for Adverse Events (CTCAE V4.0)
Acute Quality of Life changes | 0-3 months
  Expanded Prostate Cancer Index (EPIC)
Acute lower urinary symptoms | 0-3 months
  International Prostate Symptoms Score
Biochemical disease free survival | 60 months
  PSA < 0.4 ng/ml at 60 months
Number of participants with site of recurrence on mpMRI improved from PiRADS 4 or 5 to PiRADS 3 or less. | 2 years
  Number of participants with site of recurrence on mpMRI improved from PiRADS 4 or 5 to PiRADS 3 or less. If assessed by PSMA PET scan, SUV of site of disease reduced to < 3.5.

CONTACTS AND LOCATIONS:
Overall Officials: Mira Keyes, MD, Study Director — BCCA
Locations (1):
- BCCA Center for the Southern Interior, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arrayeh E, Westphalen AC, Kurhanewicz J, Roach M 3rd, Jung AJ, Carroll PR, Coakley FV. Does local recurrence of prostate cancer after radiation therapy occur at the site of primary tumor? Results of a longitudinal MRI and MRSI study. Int J Radiat Oncol Biol Phys. 2012 Apr 1;82(5):e787-93. doi: 10.1016/j.ijrobp.2011.11.030. Epub 2012 Feb 11. PMID 22331003
- [Background] Banerjee R, Park SJ, Anderson E, Demanes DJ, Wang J, Kamrava M. From whole gland to hemigland to ultra-focal high-dose-rate prostate brachytherapy: A dosimetric analysis. Brachytherapy. 2015 May-Jun;14(3):366-72. doi: 10.1016/j.brachy.2014.12.007. Epub 2015 Feb 10. PMID 25680768
- [Background] Crook J, Ots A, Gaztanaga M, Schmid M, Araujo C, Hilts M, Batchelar D, Parker B, Bachand F, Milette MP. Ultrasound-planned high-dose-rate prostate brachytherapy: dose painting to the dominant intraprostatic lesion. Brachytherapy. 2014 Sep-Oct;13(5):433-41. doi: 10.1016/j.brachy.2014.05.006. Epub 2014 Jun 20. PMID 24958556
- [Background] Da Rosa MR, Milot L, Sugar L, Vesprini D, Chung H, Loblaw A, Pond GR, Klotz L, Haider MA. A prospective comparison of MRI-US fused targeted biopsy versus systematic ultrasound-guided biopsy for detecting clinically significant prostate cancer in patients on active surveillance. J Magn Reson Imaging. 2015 Jan;41(1):220-5. doi: 10.1002/jmri.24710. Epub 2014 Jul 21. PMID 25044935
- [Background] Mason J, Al-Qaisieh B, Bownes P, Thwaites D, Henry A. Dosimetry modeling for focal high-dose-rate prostate brachytherapy. Brachytherapy. 2014 Nov-Dec;13(6):611-7. doi: 10.1016/j.brachy.2014.06.007. Epub 2014 Jul 29. PMID 25085456
- [Background] Rose JN, Crook JM, Pickles T, Keyes M, Morris WJ. Salvage low-dose-rate permanent seed brachytherapy for locally recurrent prostate cancer: Association between dose and late toxicity. Brachytherapy. 2015 May-Jun;14(3):342-9. doi: 10.1016/j.brachy.2015.01.002. Epub 2015 Feb 26. PMID 25727178